CLINICAL TRIAL: NCT03508505
Title: Postcardiotomy Venoarterial Extracorporeal Membrane Oxygenation
Acronym: PC-ECMO
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Turku University Hospital (Other Government)
Collaborators: Karolinska Institutet (Other); Ospedali Riuniti Trieste (Other); Universitätsklinikum Hamburg-Eppendorf (Other); University of Burgundy (Other); CHU de Reims (Other); Rennes University Hospital (Other); Henri Mondor University Hospital (Other); Glenfield Hospital (Other); IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other); University Hospital Muenster (Other); Institute for Clinical and Experimental Medicine (Other Government); Medical University of Vienna (Other); University Hospital, Udine, Italy (Other); Golden Jubilee National Hospital (Other Government); Heinrich-Heine University, Duesseldorf (Other); Helsinki University Central Hospital (Other); Helios Research Center (Other); Sahlgrenska University Hospital (Other); Lund University Hospital (Other); Prince Sultan Cardiac Center, Adult Cardiology Department. (Other)
Responsible Party: Sponsor
Other Study IDs: T3/2018
Record Dates: First submitted 2018-03-06; First posted 2018-04-25 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Acute Heart Failure; Low Output Heart Failure; Cardiac Output, Low; Extracorporeal Membrane Oxygenation; Cardiac Surgery; Venoarterial Extracorporeal Membrane Oxygenation
Keywords: Acute Heart Failure; Low Output Heart Failure; Cardiac Low Output; Extracorporeal Membrane Oxygenation; ECMO; Venoarterial Extracorporeal membrane oxygenation; Cardiac Surgery
MeSH Terms: conditions — Cardiac Output, Low | interventions — Extracorporeal Membrane Oxygenation; Cardiac Surgical Procedures; Coronary Artery Bypass; Transcatheter Aortic Valve Replacement; Mitral Valve Annuloplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Venoarterial extracorporeal oxygenation — Veno-arterial extracorporeal oxygenation (VA-ECMO) is inserted in the acute setting in case of cardiac low output after adult cardiac surgery in order to provide cardiopulmonary support to recovery or as bridge to transplantation.
  Other Names: Cardiac surgery; Coronary artery bypass grafting; Aortic valve replacement; Mitral valve repair; Aortic surgery

SUMMARY:
Cardiac surgery can be not infrequently complicated by cardiac low-output syndrome due to critical preoperative conditions such as cardiogenic shock, poor left ventricular function and severe myocardial ischemia. Suboptimal myocardial protection, technical errors at graft anastomoses or of prosthesis implantation, and hibernating myocardium may further contribute to cardiac low-output syndrome occurring immediately or shortly after cardiac surgery. In this setting, veno-arterial extracorporeal oxygenation (VA-ECMO) is the only means to provide cardiopulmonary support to recovery or as bridge to transplantation.

Data on the real benefit of VA-ECMO after cardiac surgery is limited and often derived from heterogeneous patient populations, which prevent conclusive results on the benefits of VA-ECMO in this setting. This issue will be investigated in the present retrospective European multicenter study.

In this setting, veno-arterial extracorporeal oxygenation (VA-ECMO) is the only means to provide cardiopulmonary support to recovery or as bridge to transplantation.

Data on the real benefit of VA-ECMO after cardiac surgery is limited and often derived from heterogeneous populations of patients who underwent different cardiac procedures. Patients with cardiac low-output after surgery for aortic dissection or valve surgery are expected to have different baseline characteristics (such as age and comorbidities) and underlying cardiac disease than patients undergoing isolated coronary surgery. Furthermore, available studies included patients operated two decades ago and this does not provide an exact measure of the benefits of this treatment strategy.

The possible benefits of using VA-ECMO after adult cardiac surgery will be investigated in this retrospective European multicenter study.

DETAILED DESCRIPTION:
Cardiac surgery can be not infrequently complicated by cardiac low-output syndrome due to critical preoperative conditions such as cardiogenic shock, poor left ventricular function and severe myocardial ischemia. Prolonged aortic cross-clamping, ischemia-reperfusion injury, suboptimal myocardial protection, technical errors at graft anastomoses or of prosthesis implantation, and hibernating myocardium may further contribute to cardiac low-output syndrome occurring immediately or shortly after cardiac surgery. In this setting, veno-arterial extracorporeal oxygenation (VA-ECMO) is the only means to provide cardiopulmonary support to recovery or as bridge to transplantation.

Data on the real benefit of VA-ECMO after cardiac surgery is limited and often derived from heterogeneous and small size series of patients who underwent different cardiac surgery procedures. Patients with cardiac low-output after surgery for aortic dissection or valve surgery are expected to have different baseline characteristics (such as age and comorbidities) and underlying cardiac disease than patients undergoing isolated coronary surgery. Furthermore, available studies included patients operated two decades ago and, in view of the development of perfusion technology and perioperative care, this does not provide an exact measure of the current benefits of this treatment strategy. Importantly, the role of intra-aortic balloon pump, left ventricular venting, duration of VA-ECMO and hospital experience should be evaluated. The investigators sought to investigate these issues in a large multicenter study.

Patients and methods Patients who were treated with VA-ECMO for cardiac low-output after adult cardiac surgery (other than heart transplantation and/or implantation of a left ventricular assist device) in 21 centers of cardiac surgery from January 2010 to December 2017.

Eligibility criteria

* Patients aged > 18 years;
* Patients who required VA-ECMO after elective, urgent or emergency adult cardiac surgery such as coronary surgery, heart valve surgery and/or aortic root surgery because of postoperative low-cardiac output syndrome and/or acute respiratory failure.

Exclusion criteria

* Patients aged < 18 years;
* Any VA-ECMO implanted before index surgical procedure;
* Patients who underwent postoperatively veno-venous ECMO;
* Patients who required VA-ECMO after heart transplantation;
* Patients who required VA-ECMO after any left ventricular assist device.

Definition criteria Definition criteria and units of measurements are reported beside each baseline, operative and postoperative variables in the electronic datasheet.

Outcomes

1. Hospital death
2. Late death
3. Stroke
4. Tracheostomy
5. Gastrointestinal complications
6. Deep sternal wound infection
7. Vascular access site infection
8. Blood stream infection
9. Peripheral vascular injury
10. Major lower limb amputation
11. New onset dialysis
12. Peak postoperative serum creatinine level
13. Nadir postoperative pH during VA-ECMO
14. Peak postoperative arterial lactate level
15. Nadir postoperative hemoglobin level
16. Chest drainage output 24 h after surgery
17. Number of red blood cells units transfused intra- and postoperatively
18. Reoperation for intrathoracic bleeding
19. Reoperation for peripheral cannulation-related bleeding
20. Intensive care unit length of stay
21. Death on VA-ECMO

Analysis of clinical results

The aim of this registry is to perform a number of analysis evaluating:

1. Early and late survival of postcardiotomy VA-ECMO;
2. Predictors and causes of in-hospital death after successful weaning from postcardiotomy VA-ECMO;
3. Comparative analysis of peripheral versus central postcardiotomy VA-ECMO;
4. VA-ECMO plus intra-aortic baloon pump vs. isolated VA-ECMO;
5. Determinants of outcome after prolonged postcardiotomy VA-ECMO (>5 days).

Publication of results The results of these studies will be submitted for publication to international, peer-reviewed journals in the fields of critical care, cardiology or cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who required VA-ECMO after elective, urgent or emergency adult cardiac surgery such as coronary surgery, heart valve surgery and/or aortic root surgery.

Exclusion Criteria:

* Any VA-ECMO implanted before index surgical procedure;
* Patients who underwent postoperatively veno-venous ECMO;
* Patients who required VA-ECMO after heart transplantation;
* Patients who required VA-ECMO after any left ventricular assist device.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who required VA-ECMO for acute heart failure occurring during the index hopsitalization for elective, urgent or emergency adult cardiac surgery such as coronary surgery, heart valve surgery and/or aortic root surgery.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Hospital death | Up to 30 days after the index cardiac surgery
  All-cause death

SECONDARY OUTCOMES:
Late death | Up to 7-year follow-up after the index cardiac surgery
  All-cause death
Stroke | Up to 30 days after the index cardiac surgery
  Ischemic infarction or hemorrhagic injury of the brain
Tracheostomy | Up to 30 days after the index cardiac surgery
  Respiratory failure requiring tracheostomy
Gastrointestinal complications | Up to 30 days after the index cardiac surgery
  Gastrointestinal complications requiring surgical treatment
Deep sternal wound infection | Up to 30 days after the index cardiac surgery
  Deep sternal wound infection or mediastinitis
Vascular access site infection | Up to 30 days after the index cardiac surgery
  Infection secondary to any vascular access
Blood stream infection | Up to 30 days after the index cardiac surgery
  Blood stream infection detected at blood cultures
Peripheral vascular injury | Up to 30 days after the index cardiac surgery
  Any aortic and/or peripheral artery complications related to VA-ECMO
Major lower limb amputation | Up to 30 days after the index cardiac surgery
  Major lower limb amputation
New onset dialysis | Up to 30 days after the index cardiac surgery
  New onset dialysis
Peak postoperative serum creatinine level | Up to 30 days after the index cardiac surgery
  Peak postoperative serum creatinine level
Nadir postoperative pH during VA-ECMO | Up to 30 days after the index cardiac surgery
  Nadir postoperative pH during VA-ECMO
Peak postoperative arterial lactate level | Up to 30 days after the index cardiac surgery
  Peak postoperative arterial lactate level
Nadir postoperative hemoglobin level | Up to 30 days after the index cardiac surgery
  Nadir postoperative hemoglobin level
Chest drainage output 24 h after surgery | Up to 24 hours after the index cardiac surgery
  Chest drainage output 24 h after surgery
Number of red blood cells units transfused intra- and postoperatively | Up to 30 days after the index cardiac surgery
  Number of red blood cells units transfused intra- and postoperatively
Reoperation for intrathoracic bleeding | Up to 30 days after the index cardiac surgery
  Reoperation for intrathoracic bleeding
Reoperation for peripheral cannulation-related bleeding | Up to 30 days after the index cardiac surgery
  Reoperation for peripheral cannulation-related bleeding
Intensive care unit length of stay | Up to 30 days after the index cardiac surgery
  Intensive care unit length of stay
Death on VA-ECMO | Up to 30 days after the index cardiac surgery
  Death on VA-ECMO

CONTACTS AND LOCATIONS:
Locations (1):
- Heart Center, Turku University Hospital, Turku, Finland

IPD SHARING:
Plan to Share IPD: Undecided
Upon request, the investigators will ask the Ethical Committee of the participating centers for permission to share all individual participant data included in this registry with the exception of data through which the patients could be identified.

REFERENCES:
- [Derived] Biancari F, Perrotti A, Ruggieri VG, Mariscalco G, Dalen M, Dell'Aquila AM, Jonsson K, Ragnarsson S, Di Perna D, Bounader K, Gatti G, Juvonen T, Alkhamees K, Yusuff H, Loforte A, Lechiancole A, Chocron S, Pol M, Spadaccio C, Pettinari M, De Keyzer D, Fiore A, Welp H. Five-year survival after post-cardiotomy veno-arterial extracorporeal membrane oxygenation. Eur Heart J Acute Cardiovasc Care. 2021 Aug 24;10(6):595-601. doi: 10.1093/ehjacc/zuaa039. PMID 33580776
- [Derived] Mariscalco G, Fiore A, Ragnarsson S, El-Dean Z, Jonsson K, Dalen M, Fux T, Ruggieri VG, Gatti G, Juvonen T, Zipfel S, Dell'Aquila AM, Perrotti A, Bounader K, Settembre N, Loforte A, Livi U, Pol M, Spadaccio C, Pettinari M, Reichart D, Alkhamees K, Welp H, Maselli D, Lichtenberg A, Biancari F; PC-ECMO group. Venoarterial Extracorporeal Membrane Oxygenation After Surgical Repair of Type A Aortic Dissection. Am J Cardiol. 2020 Jun 15;125(12):1901-1905. doi: 10.1016/j.amjcard.2020.03.012. Epub 2020 Mar 31. PMID 32305219